CLINICAL TRIAL: NCT01475006
Title: A Phase 1 First-in-Human Study Evaluating Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of AMG 595 in Subjects With Recurrent Malignant Glioma Expressing Mutant Epidermal Growth Factor Receptor Variant III (EGFRvIII)
Brief Title: AMG 595 First-in-Human in Recurrent Gliomas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20090505
Record Dates: First submitted 2011-09-29; First posted 2011-11-21 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Advanced Malignant Glioma; Anaplastic Astrocytomas; Glioblastoma Multiforme
Keywords: Epidermal Growth Factor Receptor Variant III; EGFRvIII; Glioma; Anaplastic Astrocytomas; Glioblastoma Multiforme; Antibody drug conjugate; brain tumor
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Glioma; Brain Neoplasms | interventions — AMG 595

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part I Dose Exploration (Experimental): Pre-specified nominal doses are proposed in the dose exploration. Intermediate doses may also be used if required based on the CRM design.
  Interventions: Drug: AMG 595
- Part II Dose Expansion (Experimental): Dose selected from Part 1 dose exploration
  Interventions: Drug: AMG 595

INTERVENTIONS:
Drug: AMG 595 — AMG 595 is an antibody drug conjugate that binds to EGFRvIII.

SUMMARY:
This is an open-label, sequential dose exploration study of single agent AMG 595 administered in subjects with recurrent glioblastoma multiforme (GBM) and/or anaplastic astrocytomas (AA). The purpose of the study is to evaluate safety, tolerability, and pharmacokinetics (PK) of AMG 595, and also to evaluate the objective response rate in subjects receiving AMG 595. This study will be conducted in two parts. Part 1 will explore doses of AMG 595 in subjects with recurrent GBM and/or AA. Part 2 (dose expansion) will examine the MTD established in Part 1 in subjects with recurrent GBM.

DETAILED DESCRIPTION:
This study of AMG 595 will be conducted in two parts: Part 1 (dose exploration) and Part 2 (dose expansion). Part 1 of the study is in subjects with recurrent glioblastoma multiforme (GBM) and/or anaplastic astrocytomas (AA), and Part 2 is examining the MTD in subjects with recurrent GBM. Approximately 30-40 subjects may be enrolled in Part 1, and up to 36 subjects may be enrolled in Part 2. The dose of AMG 595 utilized in Part 2 will be dependent upon data obtained in Part 1 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky performance score > or = 70%
* Must have pathologically documented, and definitively diagnosed recurrent WHO Grade IV advanced malignant glioblastoma multiforme (Part 1 and Part 2) and/or WHO Grade III anaplastic astrocytoma (Part 1 only).
* GBM and/or AA tumors expressing EGFRvIII as assessed on archived tissue by IHC staining of sections containing a minimum of 100 evaluable tumor cells.
* Archived tumor tissue from the initial diagnosis or subsequent relapse(s) of Grade IV advanced malignant glioblastoma multiforme or Grade III anaplastic astrocytoma available for submission to central review.
* Subjects with recurrent disease (confirmed by MRI and evaluable by Macdonald criteria) at the time of first or second recurrence or progression following initial definitive therapy(s)
* QTcF ≤ 470 msec
* Hematological function, as follows: Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, Platelet count ≥ 100 x 10^9/L, Hemoglobin > 9 g/dL
* Renal function, as follows: Estimated glomerular filtration rate using the Modified Diet in Renal Disease (MDRD) equation > 45 mL/min/1.73m^2, Urinary protein quantitative value of < 30 mg/dL in urinalysis or ≤ 1+ on dipstick, unless quantitative protein is < 500 mg in a 24 hr urine sample

Exclusion Criteria:

* History of central nervous system bleeding as defined by stroke or intraocular bleed (including embolic stroke) within 6 months before enrollment.
* Evidence of acute intracranial / intratumoral hemorrhage, except for subjects with stable grade 1 hemorrhage.
* Peripheral sensory neuropathy > Grade 2.
* Clinically significant ECG changes which obscure the ability to assess the PR, QT, and QRS interval; congenital long QT syndrome.
* Recent infection requiring intravenous anti-infective treatment that was completed ≤ 14 days before enrollment.
* Received radiation therapy within 12 weeks before enrollment or has not recovered from the toxic effects of such therapy.
* For Part 1 (dose escalation): Treatment with bevacizumab or antiangiogenic therapy within 4 weeks before enrollment, or for Part 2 (dose expansion): any prior treatment with bevacizumab or antiangiogenic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-02; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Clinically significant or > or = to Grade 3 CTCAE changes in safety laboratory tests, physical exams, ECGs or vital signs | 28 Days after last subject enrolled of each cohort in Part 1 and every 10, 20 and 30 subject enrolled in part 2 (if available)
PK Parameters: Cmax, Cmin, and if feasible half life - 8 time points up to 6 weeks | 28 Days after last subject enrolled of each cohort in Part 1 and every 10, 20 and 30 subject enrolled in part 2 (if available)
Objective response in GBM tumors as assessed by Macdonald criteria | 3 years
Dose limiting toxicity used to estimate the MTD | 28 Days after last subject enrolled of each cohort in Part 1 and every 10, 20 and 30 subject enrolled in part 2 (if available)

SECONDARY OUTCOMES:
Clinical benefit rate | every 6 months
Progressive free survival | 3 years
Overall survival | 3 years
Anti-AMG 595 antibody formation | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (4):
- United States (3):
  - Research Site, Los Angeles, California
  - Research Site, Boston, Massachusetts
  - Research Site, Cincinnati, Ohio
- Research Site, Parkville, Victoria, Australia

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com